CLINICAL TRIAL: NCT00456014
Title: Biological Predictors of Response to Antidepressants
Brief Title: Pre-Treatment Positron Emission Topography Scanning for Increasing Success in Antidepressant Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Miller, assistant professor of clinical psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6351R (formerly 5206); R01MH074813 (NIH); DATR A3-NSS
Record Dates: First submitted 2007-04-02; First posted 2007-04-04 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Depression
Keywords: Major Depression; Antidepressants
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Escitalopram; Desipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 - SSRI (Experimental): Participants will receive standardized pharmacotherapy with the SSRI escitalopram over 8 weeks. Non-remitters after 8 weeks will be offered standardized pharmacotherapy with desipramine
  Interventions: Drug: Escitalopram; Drug: Desipramine

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be administered at a dose of 10 mg daily for 4 weeks. If participants have not achieved response (greater than 50 % improvement in Hamilton Depression Rating Scale) by 4 weeks, the dose will be increased to 20 mg. Remission status is determined after an 8-week trial.
  Other Names: Lexapro
Drug: Desipramine — Subsequent to escitalopram trial, non-remitters will be offered pharmacotherapy with desipramine. Desipramine will be initiated at a dose of 50 mg and titrated according to a treatment manual, with monitoring of therapeutic blood levels. Remission status is determined after an 8-week trial.
  Other Names: Norpramin

SUMMARY:
This study will use pre-treatment positron emission topography and functional magnetic resonance imaging scans of the brain to predict the most effective antidepressant treatment for people with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is characterized by a combination of symptoms that can interfere with a person's ability to work, study, sleep, eat, and enjoy activities that were once pleasurable. Studies have shown that as little as 50% to 60% of individuals with MDD may respond to the first antidepressant medication prescribed. Currently psychiatrists lack tools that allow them to select the treatment plan that is most likely to benefit a particular individual. Some of the chemical abnormalities in the brains of people with MDD are detectable on positron emission topography (PET) scans. There are distinct differences in the PET scans of people with MDD who respond to treatment with a selective serotonin reuptake inhibitor (SSRI), people with MDD who do not respond to SSRI treatment, and people who do not have MDD. This study will use pretreatment PET and functional magnetic resonance imaging (fMRI) scans of the brain to predict which antidepressants will be most effective in people with MDD. This may help to reduce the trial and error currently associated with antidepressant treatment.

We will perform pretreatment PET scans to quantify serotonin transporter (5-HTT) and serotonin 1A (5-HT1A) receptor in patients with major depressive disorder (MDD). All patients will then receive a standardized treatment protocol with a selective serotonin reuptake inhibitor (SSRI), escitalopram. If the patient does not remit, he or she will receive a selective norepinephrine reuptake inhibitor (NRI), desipramine. We hypothesize those patients with high pre and postsynaptic 5-HT1A BP and low 5-HTT BP in specific brain regions will not remit to a SSRI and will remit to a selective NRI. Finally, we will generate a predictive model of remission based on brain imaging outcome measures. Our overall goal is to reduce the trial and error associated with antidepressant treatment by using data from pre-treatment quantification of 5-HT1A receptors and 5-HTT to guide antidepressant treatment selection.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of current major depressive disorder
* Currently depressed
* Subjects must be generally healthy with no significant medical problems, anemia/blood loss, or cardiac abnormalities
* Likely to tolerate medication washout
* Capacity to provide informed consent
* Off of anti-coagulant/anti-platelet treatment for 10 days
* Willing to travel to Brookhaven for PET scanning

Exclusion Criteria:

* Current abuse of or dependence on alcohol or another substance (>6 months remission okay)
* History of other major psychiatric disorders such as bipolar, schizophrenia, schizoaffective; anorexia or bulimia in past year
* First degree family history of schizophrenia if subject is under 33
* Unable/unwilling to discontinue all psychotropic medication that affects the serotonin system
* Pregnant, breastfeeding, or planning to become pregnant during the study
* A medical contraindication to antidepressants
* Dementia
* Prior head trauma with evidence of cognitive impairment
* Well-documented failure of two or more SSRI AND tricyclic antidepressant (TCA) trials of adequate dose and duration
* Metal implants, pacemaker, metal protheses or orthodontic appliance, the presence of shrapnel
* Current past, present, or anticipated exposure to radiation
* Actively suicidal
* Lifetime history of glaucoma
* Lack of response to >2 trials of antidepressant monotherapy of adequate dose and duration
* Claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramin V. Parsey, MD, PhD, Principal Investigator — Columbia University; Jeffrey M Miller, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller JM, Hesselgrave N, Ogden RT, Zanderigo F, Oquendo MA, Mann JJ, Parsey RV. Brain serotonin 1A receptor binding as a predictor of treatment outcome in major depressive disorder. Biol Psychiatry. 2013 Nov 15;74(10):760-7. doi: 10.1016/j.biopsych.2013.03.021. Epub 2013 May 9. PMID 23664414

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September 2006 to May 2012, participants were recruited through online or print advertisements, and through referrals from neighboring outpatient clinics.
Pre-assignment Details: MDD subjects who were currently on ineffective medication trial only enrolled if they were able to tolerate a medication washout.
Groups:
- Open Standardized Treatment: Participants will take escitalopram through standardized dosing over an 8 week trial. Non-remitters will be offered entry into a second open treatment phase with standardized treatment with desipramine.
  In phase 1, participants will receive escitalopram beginning at 10mg daily for 4 weeks, increasing to 20mg if non-response at week 4 or 6. If participants experience intolerable side-effects, they will be switched to an alternative SSRI, sertraline. Non-remitters after 8 weeks may enter a second phase of standardized treatment, switching from escitalopram to desipramine, dosed by blood level according to a treatment protocol. Those with intolerable side-effects to desipramine will be switched to an alternative tricyclic antidepressant, nortriptyline.
Period: SSRI Phase
Arm/Group | Open Standardized Treatment
Started | 37
Completed | 28
Not Completed | 9
Period: Tricyclic Phase
Arm/Group | Open Standardized Treatment
Started | 4 (Only non-remitters from phase 1 were eligible for phase 2, and not all those eligible continued.)
Completed | 1
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 6 subjects who started on a TCA were also enrolled in the SSRI group (switched groups due to non-remission or side effects). We analyzed data from subjects completing either 6 or 8 weeks of SSRI treatment. Reasons remaining subjects were dropped from analysis included early withdrawal, insufficient PET data and later determination of ineligibility.
Groups:
- SSRI: The single arm of this study involves patients with current MDD who will all receive open standardized treatment with escitalopram. There are not multiple arms nor multiple patient groups.
Arm/Group | SSRI
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.35 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Remission of Depressive Symptoms
Description: Remission in this study is defined as both a ≥50% decrease in the 24-item Hamilton Depression Rating Scale (HDRS) Score and a final 24-item HDRS score <10. Remission of depressive symptoms was calculated for the 28 completers of the SSRI phase.
Time Frame: Measured at Week 8
Population: 28 of 38 participants completed the SSRI phase. Only those 28 participants were assessed for remission status.
  1 participant who is counted as a non-remitter had a spontaneous remission following his MRI.
Measure: Number; unit: participants
Groups:
- 1 - SSRI: Participants will take escitalopram.
Arm/Group | 1 - SSRI
Number analyzed (Participants) | 28
participants
  Participants achieving remission | 14
  Participants failing to achieve remission | 14

2. Secondary Outcome: Remission of Depressive Symptoms - Tricyclic Phase
Description: Participants who did not achieve remission during the SSRI phase advanced to the tricyclic phase of the study. Participants were treated with either desipramine or nortriptyline. Seven participants started the tricyclic phase. Four completed the tricyclic phase. The completers (n=4) were analyzed for remission status.
Time Frame: Measured over 8 weeks
Population: Depressed participants who did not remit during the SSRI phase advanced to the tricyclic phase of the study. Five participants started treatment with desipramine, one of which also had a trial with nortriptyline. Two participants started tricyclic treatment with nortriptyline.
Measure: Number; unit: participants
Groups:
- Tricyclic Group: 7 participants who did not remit during the SSRI phase advanced to the tricyclic phase. 4 participants completed this phase.
Arm/Group | Tricyclic Group
Number analyzed (Participants) | 4
participants
  Number Achieving Remission | 1
  Numbering Failing to Remit | 3

3. Secondary Outcome: Improvement in Scores on the Hamilton Depression Rating Scale - SSRI Phase
Description: Mean % improvement from baseline to end of treatment trial using the 24-item Hamilton Depression Rating Scale. Percent improvement of depressive symptoms was calculated for the 28 completers of the SSRI phase. The higher the score on the 24-item HDRS, the greater the depression severity. Minimum score on the scale is 0, and maximum score is 74. Subscales are not used for this analysis.
Time Frame: Measured at Week 8
Population: Percent improvement of depressive symptoms was calculated for the 28 completers of the SSRI phase. 25 of the 28 SSRI participants completed a trial of escitalopram. 3 of 28 SSRI participants had intolerable side-effects to escitalopram, and were therefore switched to sertraline, and completed a trial of sertraline instead.
Measure: Mean (Standard Deviation); unit: % improvement in depression symptoms
Groups:
- 1 - SSRI: Participants will complete an 8-week trial of the SSRI escitalopram, or, if not tolerated, an 8-week trial of the SSRI sertraline.
Arm/Group | 1 - SSRI
Number analyzed (Participants) | 28
% improvement in depression symptoms
  Escitalopram Improvement | 45.46 (55.95)
  Sertraline Improvement: number analyzed (Participants) | 3
  Sertraline Improvement | 30.01 (21.87)

ADVERSE EVENTS:
Description: Systematic assessment included structured assessment using clinical global impression (CGI) therapeutic effects item at each treatment visit as well as questions regarding tolerability and side-effects of treatment intervention at each treatment visit.
Arm/Group | 1 - SSRI
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

LIMITATIONS AND CAVEATS:
small sample size, homogeneity of sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No